CLINICAL TRIAL: NCT02835222
Title: An Investigator-Sponsored Randomized Phase II Study of Selinexor in Combination With Induction/Consolidation Therapy in Acute Myeloid Leukemia Patients
Brief Title: Selinexor With Combination With Induction/Consolidation Therapy in Acute Myeloid Leukemia Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00039092; NCI-2016-00951 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 22316 (Other: Comprehensive Cancer Center of Wake Forest University); P30CA012197 (NIH)
Record Dates: First submitted 2016-07-07; First posted 2016-07-18 (Estimated); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Untreated Adult Acute Myeloid Leukemia
MeSH Terms: interventions — Cytarabine; Daunorubicin; selinexor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 2 (Selinexor) cytarabine, daunorubicin and selinexor (Experimental): INDUCTION: Cytarabine IV on days 1-7, daunorubicin hydrochloride IV on days 1-3, and selinexor PO twice weekly from day 1. Treatment continues for 14 days in the absence of disease progression or unacceptable toxicity.
  RE-INDUCTION: Disease has not responded receive cytarabine IV on days 1-5, daunorubicin hydrochloride IV on days 1-2, and selinexor PO twice weekly. Treatment continues for 14 days in the absence of disease progression or unacceptable toxicity.
  CONSOLIDATION: In remission receive cytarabine IV every 12 hours for a total 6 doses days 1-3, and selinexor PO twice weekly from day 1. Treatment repeats every 42 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cytarabine; Drug: Daunorubicin Hydrochloride; Drug: Selinexor
- Standard of Care - Cytarabine and daunorubicin (Active Comparator): INDUCTION: Cytarabine IV on days 1-7, daunorubicin hydrochloride IV on days 1-3. Treatment continues for 14 days in the absence of disease progression or unacceptable toxicity.
  RE-INDUCTION: Disease has not responded receive cytarabine IV on days 1-5, daunorubicin hydrochloride IV on days 1-2. Treatment continues for 14 days in the absence of disease progression or unacceptable toxicity.
  CONSOLIDATION: In remission receive cytarabine IV every 12 hours for a total 6 doses days 1-3. Treatment repeats every 42 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cytarabine; Drug: Daunorubicin Hydrochloride

INTERVENTIONS:
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosar-U; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Daunorubicin Hydrochloride — Given IV
  Other Names: Cerubidin; Cerubidine; Cloridrato de Daunorubicina; Daunoblastin; Daunoblastina; Daunoblastine; Daunomycin Hydrochloride; Daunomycin, hydrochloride; Daunorubicin.HCl; Daunorubicini Hydrochloridum; FI-6339; Ondena; RP-13057; Rubidomycin Hydrochloride; Rubilem
Drug: Selinexor — Given PO
  Other Names: CRM1 Nuclear Export Inhibitor KPT-330; KPT-330; Selective Inhibitor of Nuclear Export KPT-330; SINE KPT-330
  Arms: Arm 2 (Selinexor) cytarabine, daunorubicin and selinexor

SUMMARY:
This pilot phase II trial studies how well selinexor works when given together with induction, consolidation, and maintenance therapy in treating older patients with acute myeloid leukemia. Selinexor may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as cytarabine and daunorubicin hydrochloride, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Selinexor with induction, consolidation, and maintenance therapy may kill more cancer cells in older patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the overall survival of patients receiving the proposed study regimen versus standard of care (defined as time from randomization to death from any cause).

SECONDARY OBJECTIVES:

I. To compare the response rate (Complete remission (CR), complete remission with incomplete count recovery (CRi) as per Dhoner et. al.) of patients receiving the proposed study regimen versus standard of care (SOC).

II To compare disease free survival in patients receiving the proposed study regimen vs standard of care (defined as time from randomization to relapse or death from any cause).

III. To assess the rate of allogeneic stem cell transplantation

IV. To compare the toxicity of the proposed study regimen vs standard of care.

OUTLINE:

INDUCTION THERAPY: Patients receive cytarabine intravenously (IV) on days 1-7, daunorubicin hydrochloride IV on days 1-3, and selinexor orally (PO) twice weekly from day 1. Treatment continues for 14 days in the absence of disease progression or unacceptable toxicity.

RE-INDUCTION THERAPY: Patients whose disease has not responded receive cytarabine IV on days 1-5, daunorubicin hydrochloride IV on days 1-2, and selinexor PO twice weekly. Treatment continues for 14 days in the absence of disease progression or unacceptable toxicity.

CONSOLIDATION THERAPY: Patients in remission receive cytarabine IV every 12 hours on days 1-3, and selinexor PO twice weekly from day 1. Treatment repeats every 42 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 14 days and then every 3 months for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically documented newly diagnosed de novo Acute Myeloid Leukemia (non-APL) that has not yet been treated. Hydrea,cytarabine and ATRA previous treatments are acceptable.
* Patients with core binding factor acute myeloid leukemia (AML) (ie AML with t(8;21) or t(16;16) or i16) are not eligible.
* Patients must not have a secondary AML (defined as a history of prior radiation therapy or systemic chemotherapy, CMML or MDS not treated with a hypomethylating agent) however history of previous MDS treated with a hypomethylating agent IS allowed.
* Patients with de novo AML must not have partial or total monosomy 5 or 7 or i(17q) or t(17p). Negative FISH studies are sufficient for enrollment (i.e. FISH for -5, -7, +8, inv(16), t(8;21) and 17p).
* Patients must not have mutated FLT3 (either ITD OR TKD mutations).
* Hydroxyurea, leukapheresis or cytarabine may be used to control leukocytosis, provided that it is without Grade >2 non-hematologic toxicity, and can be taken until start of therapy.
* Age >18 years.
* ECOG performance status of ≤ 2 and fit for induction therapy in the opinion of the treating physician.
* Laboratory values ≤2 weeks must be:
* AST(SGOT)/ALT(SGPT)≤ 2.5 X institutional upper limit of normal
* Bilirubin ≤ 2 X ULN (3X if known history of Gilbert'syndrome)
* Creatinine clearance (CrCl) must be > 20 mL/min
* Baseline left ventricular ejection fraction of at least 40% by MUGA or ECHO.
* Female patients of childbearing potential must agree to use 2 methods of contraception (including 1 highly effective and 1 effective method of contraception) and have a negative serum pregnancy test at Screening. Male patients must use an effective barrier method of contraception if sexually active with a female of childbearing potential. For both male and female patients, effective methods of contraception must be used throughout the study and for 3 months following the last dose of study treatment.
* Ability to understand and the willingness to sign an IRB-approved informed consent document.

Exclusion Criteria:

* Patients who have received any therapy other than hydroxyurea, cytarabine or ATRA with the purpose of treating their AML or patients with core binding factor AML or Acute Promyelocytic Leukemia are not eligible.
* Patients with a secondary AML (defined as a history of prior radiation therapy or systemic chemotherapy, CMML or MDS not treated with a hypomethylating agent) however history of previous MDS treated with a hypomethylating agent IS allowed.
* Patients having received prior radiotherapy, treatment with cytotoxic agents, treatment with biologic agents or any anti-cancer therapy for a non-AML malignancy within the 4 weeks prior to treatment with selinexor, or those who have not fully recovered from the acute, non-hematological, non-infectious toxicities of any prior treatment with cytotoxic drugs, radiotherapy or other anti-cancer modalities (returned to baseline status as noted before most recent treatment).
* Patients with another active malignancy that requires treatment excluding non-melanoma skin cancers.
* Patients that have received a chemotherapy regimen with stem cell support in the previous 6 months.
* Patients with known central nervous system involvement should be excluded from this clinical trial because the penetration of selinexor into the CNS is not currently known.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to selinexor.
* Uncontrolled concurrent illness including, but not limited to symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia
* Psychiatric illness/social situations that would limit compliance with study requirements.
* Patients with known HIV infection or hepatitis (Note: Patients with known HIV infection are excluded because patients with an immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy.
* Pregnant women are excluded from this study because of the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother, breastfeeding should be discontinued.
* Patients unable to swallow tablets, patients with malabsorption syndrome, or any other GI disease or GI dysfunction that could interfere with absorption of study treatment
* Prior exposure to a SINE compound

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2018-02-02 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Overall survival | Up to 1 year
  Kaplan-Meier estimation will be used to analyze the overall survival. Overall survival (OS) is measured from the date of randomization to the date of death due to any cause. Participants will be monitored for survival through routine follow-up visits.

SECONDARY OUTCOMES:
Response rate of complete remission (CR) or complete remission with incomplete recovery (CRi) | Up to 1 year
  Confidence intervals will be calculated around the estimates of the response rate (complete remission and complete remission with incomplete recovery).
  Complete remission (CR): Defined by the absence of leukemia cells in the blood and bone marrow.
  Partial remission with incomplete hematologic recovery (CRi): This is a more stringent criterion, requiring a normal platelet count along with a normal ANC.
Progression-free survival | Up to 1 year
  Kaplan-Meier survival analysis methods to compare time to progression.
Rate of allogeneic stem cell transplantation | Up to 1 year
  Fisher's exact tests to compare rates.
Incidence of adverse events assessed by Common Terminology Criteria for Adverse Events version 4.0 | Up to 1 year
  The frequency of toxicities experienced by the participants will be presented by type and grade in an effort to monitor and report safety of the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Pardee, Principal Investigator — Wake Forest University Health Sciences
Locations (2):
- United States (2):
  - Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia